CLINICAL TRIAL: NCT02469480
Title: Intravenous Ferric Carboxymaltose vs. Oral Iron Substitution in Patients With Metastatic Colorectal Cancer (CRC) and Iron Deficiency Anemia: a Randomized Multicenter Treatment Optimization Study.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FERINJECT
Record Dates: First submitted 2015-05-13; First posted 2015-06-11 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: MCRC; iron substitution; iron deficiency anemia
MeSH Terms: conditions — Colorectal Neoplasms; Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; ferroglycine sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FERRIC CARBOXYMALTOSE (Experimental): max. 2.000 mg of ferric carboxymaltose over max. 2 weeks (max. 1.000 mg per week).
  Interventions: Drug: FerInject
- ferro sanol(R) duodenal 100 mg (Active Comparator): 200 mg ferro sanol per day over 12 weeks
  Interventions: Drug: Ferro sanol

INTERVENTIONS:
Drug: FerInject — FerInject: max. 2.000 mg of ferric carboxymaltose over max. 2 weeks (max. 1.000 mg per week).
  Arms: FERRIC CARBOXYMALTOSE
Drug: Ferro sanol — 200 mg ferro sanol per day over 12 weeks
  Arms: ferro sanol(R) duodenal 100 mg

SUMMARY:
Iron deficiency has a high prevalence in colorectal cancer patients ranging at ca. 60%. About 70% of these patients suffer from iron deficiency anemia (IDA) which adds both physical and cognitive impediments to an already straining chemotherapy. Moreover, a chronic disease like cancer often results in a reduced availability of iron for the body. In clinical practice iron substitution is usually administered orally. Due to low resorption rates, frequent gastric side effects and thus poor patient compliance a parenteral substitution seems to be a better option in terms of efficacy. In the framework of a randomized multicenter clinical trial ('FerInject') a comparison of efficacy parameters of parenteral vs. oral iron substitution will now be conducted in order to identify the best treatment form for clinical practice in oncology. Furthermore detailed quality of life-data (QoL) will be collected in both treatment arms for effect comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic or inoperable colorectal carcinoma. No curative therapy available.
2. Current palliative chemotherapy. Patients under conversion therapy must not be enrolled to this study.
3. Iron deficiency anemia: hemoglobin ≤ 10.5 g/dl and transferrin saturation < 20 % and/or serum ferritin < 20 ng/ml
4. Male and female patients aged ≥ 18 years; maturity
5. ECOG ≤ 2
6. Written informed consent
7. Life expectancy > 6 months
8. Body weight ≥ 40 kg

Exclusion Criteria:

1. Oral or intravenous iron substitution within the last 4 weeks
2. Age < 18 years or body weight < 40 kg
3. Absorption dysfunction due to short bowel syndrome or after gastric resection
4. Therapy with recombinant erythropoietin within the last 4 weeks
5. Chronic diarrhea
6. Chronic inflammatory bowel disease
7. Ferritin > 800 mg/dl at baseline
8. Hypersensitivity or contraindication to ferric carboxymaltose or iron (II) glycine sulphate complex
9. Known vitamin B12 or folic acid anemia
10. Necessary total parenteral nutrition
11. Participation in another interventional study
12. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Rise or normalization of hemoglobin | 12 weeks

SECONDARY OUTCOMES:
Fatigue as measured by EORTC-QLQ-FA13 | 12 weeks
Quality of life as measured by EORTC-C30 | 12 weeks
Handgrip strength as measured by Hydraulic Hand Dynamometer | 12 weeks
Number of allogenic blood transfusions (in total and per patient) | 12 weeks
Time until rise or normalisation of hemoglobin | 12 weeks
Genesis of the iron deficiency anemia | 12 weeks
Number of therapy with recombinant erythropoietin | 12 weeks
Dose of therapy with recombinant erythropoietin | 12 weeks
Duration of therapy with recombinant erythropoietin | 12 weeks
Inflammatory parameters | 12 weeks
Influence nutritional status on iron deficiency anemia as measured by Nutritional Risk Screening (NRS 2002) | 12 weeks
Influence nutritional status on therapy success as measured by Nutritional Risk Screening (NRS 2002) | 12 weeks
Tolerance | 12 weeks
Incidence and severity of adverse events | 12 weeks
  incidence and severity of adverse events according to CTCAE (Common Terminology Criteria for Adverse Events) Version 4 criteria as assessed at day 1, 8, 15, 36, 50 and 64 and at end of treatment.
Dropout rate due to toxicity or patient will | 12 weeks
Overall survival | 12 weeks

CONTACTS AND LOCATIONS:
Locations (18):
- Germany (18):
  - Krankenhaus Nordwest gGmbH - Institut of Clinical Cancer Research, Frankfurt am Main, Hesse
  - Klinikum Aschaffenburg, Aschaffenburg
  - Klinikum Bayreuth, Bayreuth
  - Augusta-Krankenanstalt gGmbH, Bochum
  - Medizinische Universitaetsklinik Bochum, Bochum
  - Krankenhaus Dresden-Friedrichstadt, Dresden
  - Universitätsklinikum Dresden, Dresden
  - Kliniken Essen Mitte, Essen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinik Halle-Wittenberg, Halle
  - Universitätskrankenhaus Eppendorf, Hamburg
  - NCT Heidelberg, Heidelberg
  - Gemeinschaftsklinikum Mittelrhein GmbH, Koblenz
  - Universitätsmedizin Mannheim, Mannheim
  - Klinikum rechts der Isar, Munich
  - Klinikum Bogenhausen, Munich
  - Elblandklinikum Riesa, Riesa
  - Caritas Klinikum St. Theresia, Saarbrücken

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- See also: Related Info — http://www.ikf-nordwest.de/home-studien.html?study=156